CLINICAL TRIAL: NCT05027711
Title: Magnetic Resonance-guided Adaptive Stereotactic Body Radiotherapy for Hepatic Metastases - MAESTRO -
Brief Title: Magnetic Resonance-guided Adaptive Stereotactic Body Radiotherapy for Hepatic Metastases
Acronym: MAESTRO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Juergen Debus, Department Head, University Hospital Heidelberg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RADONK-MAESTRO-2020
Record Dates: First submitted 2021-08-03; First posted 2021-08-30 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Hepatic Metastasis
Keywords: Magentic Resonance-guided Adaptive Stereotactic Body Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Experimental): Magnetic Resonance-guided Stereotactic Body Radiotherapy (MRgSBRT), if a biologically effective dose (BED) of ≥ 100 Gy is achievable using an ITV
  Interventions: Radiation: MRgSBRT (Magnetic Resonance-guided Stereotactic Body Radiotherapy)
- B (Experimental): ITV (Internal target volume)-based Stereotactic Body Radiotherapy (ITV-SBRT), if a biologically effective dose (BED) of ≥ 100 Gy is achievable using an ITV
  Interventions: Radiation: ITV (Internal target volume)-based Stereotactic Body Radiotherapy (ITV-SBRT)
- C (Experimental): Magnetic Resonance-guided Stereotactic Body Radiotherapy (MRgSBRT). If a BED of ≥ 100 Gy cannot be achieved using an ITV concept (e.g. due to OAR constraints), patients will be treated in arm C using MRgSBRT with the highest achievable dose as deemed appropriate by the treating radiation oncologist
  Interventions: Radiation: MRgSBRT (Magnetic Resonance-guided Stereotactic Body Radiotherapy)

INTERVENTIONS:
Radiation: ITV (Internal target volume)-based Stereotactic Body Radiotherapy (ITV-SBRT) — ITV (Internal target volume)-based Stereotactic Body Radiotherapy (ITV-SBRT)
  Arms: B
Radiation: MRgSBRT (Magnetic Resonance-guided Stereotactic Body Radiotherapy) — MRgSBRT (Magnetic Resonance-guided Stereotactic Body Radiotherapy)
  Arms: A; C

SUMMARY:
Stereotactic body radiotherapy (SBRT) is an established local treatment method for patients with hepatic oligometastases. Liver metastases often occur in close proximity to radiosensitive organs at risk (OARs). This limits the possibility to apply sufficiently high doses needed for optimal local control. MR-guided radiotherapy (MRgRT) is expected to hold potential to improve hepatic SBRT by offering superior soft-tissue contrast for enhanced target identification as well as the benefit of daily real-time adaptive treatment. The MAESTRO trial therefore aims to assess the potential advantages of adaptive, gated MR-guided SBRT (MRgSBRT) compared to conventional SBRT at a standard linac using an ITV (internal target volume) approach (ITV-SBRT).

DETAILED DESCRIPTION:
Hepatic SBRT is a well-established local treatment method for technically or medically inoperable hepatic metastases. However, clinicians are often restricted in the utilization of hepatic SBRT due to dose limitations of the uninvolved liver and nearby OARs (e.g. small bowel, stomach, kidney). MR-guided radiotherapy with its superior soft-tissue contrast is believed to facilitate the precise detection of tumor position and interfractional changes in patient anatomy. Respiratory gating at the MR-Linac enables real-time visualization of the tumor as well as synchronization of beam delivery to the patient's breathing . Therefore, safety margins and thus the irradiated volume can possibly be decreased with MRgSBRT in comparison to ITV-based SBRT, reducing the risk of treatment-associated toxicity. Hepatic MRgSBRT of smaller target volumes might further offer the possibility of dose escalation for increasing local control. To our knowledge, only two retrospective analyses including 26 and 29 patients as well as one case report about hepatic MR-guided SBRT using a MR-Linac can be found in literature. As MR-guided adaptive SBRT is very staff intense and time consuming compared to standard ITV-based SBRT, prospective studies are needed to demonstrate the expected benefits of MR-guided adaptive SBRT. This trial will be conducted as a prospective, randomized, three-armed phase II study in 82 patients with hepatic metastases (solid malignant tumor, 1-3 hepatic metastases confirmed by magnetic resonance imaging (MRI), maximum diameter of each metastasis ≤ 5 cm (in case of 3 metastases: sum of diameters ≤ 12cm), age ≥ 18 years, Karnofsky Performance Score ≥ 60%). If a biologically effective dose (BED) ≥ 100 Gy is feasible based on ITV-based planning, patients will be randomized to either MRgSBRT (Arm A) or ITV-based SBRT (Arm B). If a lesion cannot be treated with a BED ≥ 100 Gy, the patient will be treated in Arm C with MRgSBRT at the highest possible dose.

ELIGIBILITY:
Inclusion Criteria:

* confirmed underlying solid malignant tumor (no germ cell tumor, leukemia, lymphoma)
* 1-3 hepatic metastases confirmed by pre-therapeutic MRI
* indication for SBRT of 1-3 hepatic metastases
* maximum diameter each hepatic metastasis ≤ 5 cm (in case of 3 metastases: sum of diameters ≤ 12 cm)
* age ≥ 18 years of age
* Karnofsky Performance Score ≥ 60%
* ability to lie still on the radiotherapy treatment couch for at least one hour
* ability to hold one's breath for more than 25 seconds
* for women with childbearing potential, adequate contraception
* ability of subject to understand character and individual consequences of the clinical trial
* written informed consent (must be available before enrolment in the trial)

Exclusion Criteria:

* refusal of the patients to take part in the study
* patients with primary liver cancer (eg. HCC, CCC)
* patients after liver transplantation
* impairment of liver function to an extent contraindicating radiotherapy (to the discretion of the treating radiation oncologist)
* active acute hepatic/biliary infection (e.g. hepatitis, cholangitis, cholecystitis)
* previous radiotherapy of the hepatobiliary system, if previous and current target volumes overlap MAESTRO Study Studienprotokoll Seite 25 von 54 Version 1.0 vom 17.12.2020
* patients who have not yet recovered from acute toxicities of prior therapies
* claustrophobia
* pregnant or lactating women
* contraindications against performing contrast-enhanced MRI scans (pacemakers, other implants making MRI impossible, allergy to gadolinium (GD)-based contrast agent)
* participation in another competing clinical study or observation period of competing trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-08-12 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Treatment related Toxicity | within the first year after radiation treatment
  occurrence of treatment-related gastrointestinal or hepatobiliary CTCAE V5.0 toxicity of grade III or higher

SECONDARY OUTCOMES:
Treatment related Toxicity | within 24 months after radiation treatment
  assesment of toxicity according to CTCAE V5.0 in all three treatment groups
Treatment related Quality of life | within 24 months after radiation treatment
  Changes in quality of life according to EORTC QLQ C-30
Treatment related Quality of life | within 24 months after radiation treatment
  Changes in quality of life according to EORTC QLQ LMC-21
local Tumor Control | within 24 months after radiation treatment
  Change of local Tumor size at one specific site
locoregional control | within 24 months after radiation treatment
  Change of local Tumor size within a defined local region
distant tumor control | within 24 months after radiation treatment
  apparence of distant Tumor leasions
progression-free survival (PFS) | 24 months after radiation treatment
  time of suvival without Tumor progression
overall survival (OS) | 24 months after radiation treatment
  time of Survival of studypopulation
Changes in applied biological effective doses (BED) to the target Volumen (Tumor) | through study completion, an average of 1 year
  BED increase and OAR doses with MRgSBRT compared to initial ITV-based planning in arms A and C
Evaluation of potential prognostic biomarkers | within 24 months after radiation treatment
  Changes in blood Levels of blood Parameters compared to reference samples

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Heidelberg, Radiation Oncology, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoegen P, Zhang KS, Tonndorf-Martini E, Weykamp F, Regnery S, Naumann P, Lang K, Ristau J, Korber SA, Dreher C, Buchele C, Rippke C, Renkamp CK, Paul KM, Konig L, Busch C, Krisam J, Sedlaczek O, Schlemmer HP, Niyazi M, Corradini S, Debus J, Kluter S, Horner-Rieber J. MR-guided adaptive versus ITV-based stereotactic body radiotherapy for hepatic metastases (MAESTRO): a randomized controlled phase II trial. Radiat Oncol. 2022 Mar 27;17(1):59. doi: 10.1186/s13014-022-02033-2. PMID 35346270